CLINICAL TRIAL: NCT02397070
Title: Effectiveness of a Jaw Exercise Program in Temporomandibular Disorders Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Wagner Araujo de Negrieiros, Wagner Araujo de Negreiros, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Federal University of Ceara
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Temporomandibular Joint Disorders; Musculoskeletal Diseases
Keywords: Jaw exercise; Occlusal splint; Treatment; Muscular pain; Mandibular movement
MeSH Terms: conditions — Temporomandibular Joint Disorders; Musculoskeletal Diseases; Myalgia | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jaw exercise program (Experimental)
  Interventions: Procedure: Jaw exercise program
- Occlusal splint and counseling (Active Comparator)
  Interventions: Device: Occlusal Splint and counseling

INTERVENTIONS:
Procedure: Jaw exercise program — The jaw exercise program will consist of three cycles: 1st CYCLE - simple opening and closing mouth, right and left lateral excursions with mechanisms of proprioceptive neuromuscular facilitation and muscle coordination; 2 ° CYCLE - opening and closing exercises, right and left lateral excursions with a counter-resistance force imposed by the participant, with reciprocal inhibition, stretching, and muscular endurance mechanisms; 3rd CYCLE - specific exercises to disk capture attempt in cases of disk displacement with reduction and acute disk displacement without reduction (mouth opening and closing in protrusion) or chronic disk displacement without reduction (forced mouth opening in order to push the disc), with remodeling articulate mechanisms. The conduct will be individualized according to the need and symptoms of patients, which will be monitored fortnightly. It will be proposed 3 times a day, lasting a minute and a half per turn, in front of the mirror, during three months.
  Arms: Jaw exercise program
Device: Occlusal Splint and counseling — The occlusal splints will be made from obtaining a plaster type IV model of upper arch using alginate and metal stock tray. A 2mm thick polyacetate blade will be adapted to the vacuum device plasticizer, heated and pressed over the previously cut U-shaped plaster model. After cooling, it will be added the self-curing acrylic resin on occlusal surface in order to increase the vertical dimension of occlusion in 2mm (anterior region). After polishing, the splints will be intraorally adjusted using carbon paper and clamp Muller, and installed obtaining maximum tooth contacts in centric relation. The splints will be flat and of full coverage for night use. Patients will be monitored every two weeks for the occlusal adjustment for three months. It will also be done counseling measures through a printed guide in relation to the daily care and the various contributing factors of TMD (diet, stress reduction, elimination of parafunctions and posture correction).
  Other Names: Occlusal appliances,; Occlusal plates
  Arms: Occlusal splint and counseling

SUMMARY:
This study evaluates the effect of jaw exercise therapy in the treatment of temporomandibular disorder patients (TMD). An eligible group of patients will be treated with that therapy (experimental group) and another group will be treated with counseling and occlusal splint (control group), considered the standard therapy for TMD.

DETAILED DESCRIPTION:
Mandibular exercises may have behavioral and cognitive action, educating the patient and serving as an instrument of control of parafunctional activity. It is a simple, easy, which seeks adherence to treatment and has negligible cost. A disadvantage is the need of motivation and discipline of the patient in carrying out the therapy daily. The occlusal splints, associated with educational guidance and counseling have world indication the possibility of promoting teeth protection, joint decompression, equalization of electromyographic activity, conscious control of parafunctional activity and strong placebo effect.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 20-45 years, clinical diagnosis of muscular TMD form mild to moderate according to the Criteria of the Diagnostic and Research of TMD (RDC / TMD), good reception and understanding of spoken Portuguese, able to provide a informed consent, and be available to attend the evaluation returns.

Exclusion Criteria:

* Rheumatic, vascular, neurological, infectious or neoplastic disease, cognitive or motor problems, pregnancy status or use of abusive drugs, chronic facial pain history (2 years or more), refuses to participate in the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Muscular pain | Three months
  Pain on masticatory muscles (masseter and temporal) pressure, scored 0-3 (0=no pain, 3= severe pain).
Articular pain | Three months
  Pain on bilateral digital pressure on articular region, scored 0-3 (0=no pain, 3= severe pain).

SECONDARY OUTCOMES:
Maximum mouth opening | Three months
  Mouth opening amplitude, measured with a millimeter ruler from the tip of the lower incisors to the tip of the upper incisors, counting the vertical crossover.
Mandibular excursions | Three months
  Lateral and protrusive movement, measured with a millimeter ruler considering the right and left lateral excursion and protrusive excursion.

CONTACTS AND LOCATIONS:
Overall Officials: Wagner A Negreiros, PhD, Principal Investigator — Universidade Federal do Ceara
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

REFERENCES:
- [Result] Kraaijenga S, van der Molen L, van Tinteren H, Hilgers F, Smeele L. Treatment of myogenic temporomandibular disorder: a prospective randomized clinical trial, comparing a mechanical stretching device (TheraBite(R)) with standard physical therapy exercise. Cranio. 2014 Jul;32(3):208-16. doi: 10.1179/0886963413Z.00000000016. Epub 2014 Jan 24. PMID 25000163
- [Result] Craane B, Dijkstra PU, Stappaerts K, De Laat A. Randomized controlled trial on physical therapy for TMJ closed lock. J Dent Res. 2012 Apr;91(4):364-9. doi: 10.1177/0022034512438275. Epub 2012 Feb 8. PMID 22318373
- [Result] Yoda T, Sakamoto I, Imai H, Honma Y, Shinjo Y, Takano A, Tsukahara H, Morita S, Miyamura J, Yoda Y, Sasaki Y, Tomizuka K, Takato T. A randomized controlled trial of therapeutic exercise for clicking due to disk anterior displacement with reduction in the temporomandibular joint. Cranio. 2003 Jan;21(1):10-6. doi: 10.1080/08869634.2003.11746226. PMID 12555926
- [Result] Yoshida H, Kashiwagi K, Sakata T, Tanaka M, Kawazoe T, Morita S. Prognostic factor of mandibular condylar movement exercise for patients with internal derangement of the temporomandibular joint on initial presentation: preliminary report. J Craniomaxillofac Surg. 2013 Jul;41(5):356-8. doi: 10.1016/j.jcms.2012.05.009. Epub 2012 Jul 11. PMID 22789869